CLINICAL TRIAL: NCT02086279
Title: AMH Levels Change During Treatment With GnRh Agonist: A Prospective Observational Study.
Brief Title: AMH Levels Change During Treatment With GnRh Agonist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMHunderGnRH
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Uterine Fibroids; Endometriosis; Endometriosis of Uterus; Pelvic Pain
Keywords: AMH levels; Ovarian reserve; GnRH analogue; Ovarian reserve after GnRH analogue; Ovarian reserve modification; Antral follicle count; Antral follicle count after GnRH analogue
MeSH Terms: conditions — Leiomyoma; Endometriosis; Adenomyosis; Pelvic Pain | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GnRH analogue (No Intervention): Patients with uterine myoma, endometriosis, fibromatous uterus, chronic pelvic pain in list for surgery are usually pharmacologically treated by administration of GnRHa, 11.25 mg at 21° day of the menstrual cycle and repeated after 3 months to reduce pain symptoms, menstrual blood loss, uterine or fibroids vascularization and size, during the months spent on surgery waiting list.
  Patients enrolled will be subjected to valuation of ovarian reserve: specifically, serum levels of AMH and antral follicle count (AFC) between 1 and 4 days of the menstrual cycle will be measured at study entry and at 1, 3 and 6 months after the administration of the first vial of GnRH-a
  Interventions: Drug: GnRH analogue

INTERVENTIONS:
Drug: GnRH analogue — Patients with uterine myoma, endometriosis, fibromatous uterus, chronic pelvic pain in list for laparoscopic surgery or laparotomy are usually pharmacologically treated by administration of GnRHa, 11.25 mg at 21° day of the menstrual cycle and repeated after 3 months. This treatment is part of our preoperative routine in order to reduce pain symptoms, menstrual blood loss, uterine or fibroids vascularization and size, during the months spent on surgery waiting list.
  Patients who will satisfy inclusion and exclusion criteria will be enrolled in this study protocol and will be subjected to valuation of ovarian reserve: specifically, serum levels of AMH and antral follicle count (AFC) between first and fourth days of the menstrual cycle will be measured.
  Other Names: Gonadotropin-releasing hormone analogue

SUMMARY:
To evaluate the variation of AMH levels in women undergoing treatment with GnRHa, and to assess whether this variation correlates with changes in the antral and pre-antral follicle ultrasonographic count (AFC).

DETAILED DESCRIPTION:
The anti Mullerian hormone (AMH) is a glycoprotein produced by granulosa cells of antral and preantral ovarian follicles.

Several studies have shown that the AMH levels provide a reliable indication of the size of the growing follicles pool (1). AMH is now commonly used as a biomarker for improving the ovarian reserve in women of reproductive age because it is related with outcomes of assisted reproduction cycles, chances of pregnancy and distance from menopause (2-4).

For several years GnRH agonists have been used for the purpose of preserving fertility in the course of chemotherapy in young women with cancer (5). Their effectiveness, however, isn't 100% and there is the need to monitor the ovarian reserve in the course of treatment in these young women. With the administration of GnRHa, the FSH levels (the most used hormone for improve the ovarian reserve, although it is less reliable and less manageable because of its intra-cyclic variations) cannot be used to measure the residual ovarian function due to the physiological reduction of gonadotropins induced by the treatment. AMH levels, conversely, are relatively stable both during the menstrual cycle (6) and during administration of the contraceptive pill (7,8), suggesting the gonadotrophin independence of this molecule. AMH could therefore be a useful biomarker of ovarian reserve in the course of GnRHa treatment.

The use of GnRHa for fertility preservation during chemotherapy is controversial because of inconclusive outcome data on fertility (9) and because the mechanism by which GnRHa may act to preserve fertility is unknown. The major function of GnRHa is to suppress the production of pituitary gonadotrophins, acting indirectly on the ovarian follicles, not exposing growing follicles to the toxicity of chemotherapy and thus protecting the future ovarian function.

Determine the effect of GnRHa on AMH serum level is an essential step to determine both the effectiveness of the treatment in terms of preservation of fertility and the reliability of this marker for ovarian reserve in cancer patients treated with GnRHa. Up to now, the published studies have shown extremely contrasting data. Considered that GnRHa is largely used in non-oncological patients for preoperative pharmacological preparation in various benign gynecological conditions, it is possible to exploit the high number of patients with these characteristics for the non-invasive assessment of analogue effect on the AMH levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients waiting for surgery for benign conditions such as uterine fibroids and endometriosis, undergoing preoperative treatment with two consecutive doses of GnRHa at a dose of 11.25 every three months
* 18 to 45 years aged patients
* Regular menstrual intervals between 22 and 35 days
* Expressed written consent for the study entry

Exclusion Criteria:

* Patients who do not consent to pharmacological preparation with GnRHa
* Estrogen-progestin therapy in the 2 months before enrollment
* Autoimmune diseases, chronic , metabolic, systemic and endocrine disorders, including hyperandrogenism, hyperprolactinemia, diabetes mellitus and thyroid disease.
* Hypogonadotropic hypogonadism
* Majors clinical conditions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
AMH levels change before and after GnRHa | At study entry and at 1, 3 and 6 months after the administration of the first vial of GnRH-a

SECONDARY OUTCOMES:
Preantral and antral follicles | At study entry and at 1, 3 and 6 months after the administration of the first vial of GnRH-a
Correlation between AMH levels and preantral and antral follicles count | At study entry and at 1,3 and 6 months after the first vial of GnRH

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy